CLINICAL TRIAL: NCT05208645
Title: The Place of Men in Arrested Pregnancies
Acronym: PHGA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8298
Record Dates: First submitted 2021-08-06; First posted 2022-01-26 (Actual); Last update posted 2022-01-26 (Actual); Status verified 2021-08

CONDITIONS: Arrested Pregnancies
Keywords: arrested pregnancies; Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An terminated pregnancy is defined as the cessation of cardiac activity before 14 weeks of amenorrhea. This early interruption of gestation can be induced by pathological, traumatic or idiopathic causes. In any case, it remains a physically and psychologically trying event for the woman, the couple as well as for the man.

Indeed, the loss of this embryo, which measures only a few millimeters, corresponds to the loss of a child for the triad: woman, man, couple. The termination of this pregnancy is experienced as a bereavement for the future parents.

The stopped pregnancy has always been a taboo in the society. The proof being that it was not until the 1980s that this was considered mourning and its psychological consequences were studied.

Following these studies, psychological follow-ups are democratized and are thus offered to women. However, when is it men? The investigators have always put the woman at the center of the care process. Which is legitimate. However, the man is often seen as "the person who influences the woman". This default categorization marginalizes the man who would like to be an actor in the care of his partner. In fact, men are increasingly asking to support women in their gynecological care procedures. Unfortunately, for lack of measures put in place. The men are more than abandoned.

ELIGIBILITY:
Inclusion criteria:

* Age ≥18 years old
* male
* Speaking French
* The progenitor of the pregnancy and whose partner is affected by an aborted pregnancy

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* Subject under safeguard of justice
* Subject under guardianship or guardianship
* Subject under guardianship, curatorship or safeguard of justice

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Male adult who is progenitor of the pregnancy and whose partner is affected by an aborted pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-31 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Identify the role of the men's place during an aborted pregnancy of their partners | up to 1 month post-arrested pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Luisa ATTALI, Midwife, Principal Investigator — Service de gynécologie Obstétrique - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de gynécologie Obstétrique - Hôpitaux Universitaires de Strasbourg, Strasbourg, France